CLINICAL TRIAL: NCT06864078
Title: Diclofenac Potassium and Lidocaine Gel in Posterior Vaginal Fornix Prior to IUCD Insertion in Patients Delivered by Cesarean Section
Brief Title: IUCD Insertion in Patients Delivered by Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Safaa Bashandy Hussein, Resident of Obstetrics & Gynecology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Safaa Bashandy
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2023-09

CONDITIONS: IUD
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Study Group) (Active Comparator): About 64 women who received lidocaine gel and diclofenac potassium tablets,to be administered 1 hour before planned intrauterine device insertion (Cu T380A) insertion, according to the assigned group. A syringe consists of six millimeters of two percent lidocaine gel (Xylocaine Jelly, AstraZeneca, Australia) for the active management group
  Interventions: Device: IUD Insertion during Cesarean Section; Drug: lidocaine gel and diclofenac potassium tablets
- Control Group (Placebo Comparator): About 64 women who received placebo tablets and placebo gel,2 placebo tablets to be administered 1 hour before planned intrauterine devices insertion (Cu T380A) insertion,six millimeter of placebo gel (K-Y jelly, Johnson & USA, Johnson).
  Interventions: Device: IUD Insertion during Cesarean Section; Drug: Placebo

INTERVENTIONS:
Device: IUD Insertion during Cesarean Section — to evaluate the analgesic effect of diclofenac potassium and lidocaine gel applied to the posterior vaginal fornix before IUD insertion in women who had previously undergone cesarean section. By assessing the efficacy of this pain management strategy, this study seeks to contribute to the optimization of IUD insertion protocols, improving patient comfort and increasing the acceptance of this highly effective contraceptive method.
Drug: lidocaine gel and diclofenac potassium tablets — lidocaine gel and diclofenac potassium tablets
  Arms: Group I (Study Group)
Drug: Placebo — Placebo
  Arms: Control Group

SUMMARY:
Long-acting reversible contraceptive (LARC) methods, including intrauterine devices (IUDs), are highly effective and safe options for preventing unintended pregnancies. IUDs have failure rates below one percent, making them one of the most reliable forms of contraception available.

They are suitable for females of all ages, including adolescents and nulliparous women, and offer long-term protection without requiring daily adherence, unlike oral contraceptives. Increasing the utilization of IUDs can provide a safe, long-acting, highly effective, and reversible method of contraception, reducing the incidence of unintended pregnancies and associated complications.

DETAILED DESCRIPTION:
One of the primary concerns for women who have undergone a C-section is the recovery time. C-sections are major surgeries, and the recovery process can be longer and more uncomfortable than that of a vaginal delivery. Women who have had a C-section may experience pain, discomfort, and fatigue for several weeks after the procedure. Additionally, they may be required to take pain medication, which can cause side effects such as nausea and drowsiness.

Women who have had a C-section may also experience emotional difficulties following the procedure. The recovery process can be difficult, and the physical limitations imposed by the surgery may make it difficult for women to care for their newborns. Additionally, some women may feel a sense of disappointment or failure if they were not able to deliver their baby vaginally.

On the other hand, vaginal delivery is considered to be less invasive than a C-section, and the recovery process is typically faster and less uncomfortable. Women who have had a vaginal delivery may be able to return to their normal activities more quickly than those who have had a C-section. Additionally, vaginal delivery allows for immediate skin-to-skin contact between the mother and baby, which can promote bonding and breastfeeding.

Another advantage of vaginal delivery is that it is associated with a lower risk of complications for both the mother and the baby. C-sections are considered to be major surgeries, and as such, they carry a higher risk of complications such as infection, bleeding, and blood clots. Additionally, babies born via C-section are at a slightly higher risk of respiratory problems and other complications.

One of the most important factors in determining the quality of life after childbirth is the woman's physical and emotional well-being. Women who have had a C-section may experience more physical discomfort and emotional distress in the immediate aftermath of the procedure. However, the long-term effects of C-sections on a woman's physical and emotional well-being are not well understood.

Despite their effectiveness, IUD insertion can be associated with significant discomfort and pain, which may deter some women from choosing this contraceptive method. Pain during IUD insertion arises from several factors, including myometrial contractions triggered by the device irritating the uterine cavity, passage through the cervical canal, and the application of a tenaculum to stabilize the cervix. The insertion process involves measuring the uterine cavity with a sound, followed by advancing the IUD through the cervix and into the uterus, all of which can stimulate pain receptors and cause discomfort.

Expulsion of an IUD occurs in approximately one in twenty women, with the highest risk during the first three months following insertion, particularly after menstruation. Proper training for healthcare providers and the use of pain management strategies can help minimize these risks and improve the overall experience for women undergoing IUD insertion.

Pharmacological interventions to alleviate pain during IUD insertion include local anesthetics, nonsteroidal anti-inflammatory drugs (NSAIDs), and prostaglandins to soften the cervix. However, there is considerable variability in the application of these strategies, with no universally accepted pain management protocol.

Diclofenac potassium is a potent, rapidly acting NSAID with well-documented analgesic properties.

The combined use of diclofenac potassium and lidocaine gel offers a dual approach to pain relief. Lidocaine gel alleviates pain originating from cervical instrumentation, such as tenaculum application and passage of the sound and IUD through the cervical canal, while diclofenac potassium mitigates pain from the uterus and cervix by inhibiting inflammatory pathways

ELIGIBILITY:
Inclusion Criteria:

* Women at term pregnancy willing to give birth at the hospital, either via c-section or vaginal delivery.- - - Singleton pregnancy with viable fetus.
* Women who are willing and able to provide informed consent to participate in the study.
* Women who are able to communicate in the language of the study, either verbally or through a translator

Exclusion Criteria:

* Women who have a medical condition that would prevent them from participating in the study, such as severe mental illness.
* Women with medical disorder during pregnancy as pre-eclampsia.
* Having a history of dystocia or instrumental delivery, stillbirth, giving birth to a child with a weight of less than 2500 grams, having a history of general medical conditions, disabilities, depression, drug intake, major psychological problems, or having stress-inducing experiences such as the loss of a family member, divorce, or family problems.
* Individuals with medical conditions such as low back pain, chronic constipation, urination problems, or breast problems before pregnancy.
* Women who have had multiple c-sections in the past.
* Women who were not able to give a birth vaginally due to medical reasons such as placenta previa, cord prolapse, or fetal distress.
* Women who are not willing or able to provide informed consent to participate in the study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Pain Management | 2 hours
  Assessing the efficacy of the pain strategy resulted from IUD insertion By using VAS scale and improving patient comfort and increasing the acceptance of this highly effective contraceptive method

CONTACTS AND LOCATIONS:
Overall Officials: Yousry Omar Salim El Maraghy, Professor, Study Chair — Obstetrics and Gynecology, Faculty of medicine Al-Azhar University Assuit.
Locations (1):
- Al-Azhar University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided